CLINICAL TRIAL: NCT00927355
Title: Effects of Thiazolidinediones on Human Bone Marrow Stromal Cell Differentiation Capacity:In Vitro and In Vivo- A Pilot Study
Brief Title: Effect of Thiazolidinediones on Human Bone
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Natasha Khazai, M.D., assistant professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: IRB00014509; 08006 (Other: Other)
Record Dates: First submitted 2009-06-24; First posted 2009-06-25 (Estimated); Results first posted 2014-06-02 (Estimated); Last update posted 2016-03-29 (Estimated); Status verified 2016-03

CONDITIONS: Osteoblast; Adipocytes; Bone Density; Osteocalcin; Adiponectin; Mesenchymal Stem Cells
Keywords: pioglitazone; human bone marrow stem cells; adipocytes; osteoblasts; bone mineral density; adiponectin; leptin; CTX; P1NP; Osteocalcin
MeSH Terms: interventions — Pioglitazone

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pioglitazone (Active Comparator): half of the diabetic patients will be randomized to pioglitazone treatment for 6 months starting out with 15mg qd for 4 weeks and dose increased to 30mg (2 tablets) qday if no adverse effects noted at the four week mark by study physician.
  Interventions: Drug: Pioglitazone
- Placebo (Placebo Comparator): The other half will be randomized to placebo for 6 months. The placebo pills also start out with one "15mg) pill qday and are increased to 2 tablets ("30mg") qday after 4 weeks if no adverse effects are noted by study physician.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pioglitazone — 6 month treatment with pioglitazone 15mg for four weeks with dose increased to 30mg if no adverse effects (swelling of lower extremities, liver enzyme elevation) noted at the four week mark.
  Other Names: Actos
  Arms: Pioglitazone
Drug: Placebo — The placebo pills also start out with one ("15mg") pill qday and are increased to 2 tablets ("30mg") qday after 4 weeks if no adverse effects are noted by study physician.
  Arms: Placebo

SUMMARY:
We will prospectively study 2 groups of diabetic patients treated with pioglitazone or placebo for 26 weeks. Bone marrow aspirates will be obtained from these patients at baseline and after 26 weeks of treatment, and hBMCs will be isolated from these bone marrow aspirations. The ability of hBMCs to differentiate into osteoblast and adipocytes lineages will be compared before and after treatment with pioglitazone and compared to placebo. In parallel, clinical markers of bone formation and resorption as well as bone mineral density will be assessed before and after 26 weeks of treatment. Primary endpoint for this study will be detection of change in number of osteoblasts or adipocytes from cultured hBMCs between study groups and within each group.

DETAILED DESCRIPTION:
E2a. Screening: Prescreening of electronic medical records will be used as much as possible to reduce screen failure rates. Patients will undergo a full history (with special focus on inclusion and exclusion criteria), physical exam, and blood draw. Lab work will consist of CBC, PT, PTT, CMP, HbA1c, PTH, serum beta-HCG in females of childbearing potential and testosterone in males. We will measure 25(OH) Vitamin D at baseline and completion of the study.

E2b. Study visits Subjects will be admitted to the Grady GCRC after an overnight fast at the initial visit and at 26 weeks. Study drug will be dispensed at the initial visit. At the initial visit and at 26 weeks, subjects will undergo bone marrow aspiration by a skilled and certified Hematology Oncology fellow, bone densitometry (DXA) of their hip and spine, and a blood.draw (5mls).

Subjects will be seen in follow-up at the Grady GCRC at 2 weeks and every 4 weeks thereafter for measurement of body weight, vital signs, and targeted history looking for any side effects from study drugs.

Study drug will be dispensed to patients at baseline and on monthly follow-up visits thereafter. To assess compliance, subjects will be instructed to return any unused drug, and if the subject takes less than 75% of the study medication, the patient will be withdrawn from the study. Patients will be monitored closely for development of side effects. Glycemic control will be assessed with HbA1c measurements at baseline, 12 weeks into the study and at end of study. Home blood sugars, fasting and occasional postprandial blood sugars will be assessed at each of the study visits.

E2b.2. Bone Marrow Biopsy aspiration: Bone marrow (BM) aspiration will be done by a hematology and oncology fellow, Dr. Simbo Aduloju, who is certified in doing these procedures at the Grady GCRC. Subjects will be pre-medicated 30 minutes prior to the procedure with oral Lorazepam 2mg and Tylenol 500mg for analgesia.The only absolute contraindication to BM aspirations is the presence of bleeding disorders. During the screening process, patients will be asked about a history of coagulopathies such as hemophilia. In addition all patients will have their PT, PTT and platelets checked at baseline. Under sterile technique and after local anesthesia with 2% lidocaine, 5mls of bone marrow will be aspirated from the posterior iliac crest using a 16 gauge bone marrow aspiration needle attached to a 10 ml syringe. The sample will be placed on ice immediately and transported to the lab of Dr. George Beck. After the procedure, manual pressure will be applied to the aspiration site for a minimum of 5 minutes to prevent bleeding. Patients blood pressure will be checked after the procedure and prior to their departure from the GCRC to ensure absence of hypotension due to lorazepam.

E2b.2.1. Please see section E2c. below for experimental design on procurement of hBMCs from bone marrow aspirates and determination of osteoblast/adipocyte differentiation capacity from these hBMCs.

E2b.3. BMD Evaluation: DXA measurements will be performed at the spine and dominant hip (contralateral hip in the presence of hardware in the dominant hip) using a GE Lunar Prodigy Instrument (GE medical Systems) at Grady Memorial Hospital. The DXA scanner is calibrated on a daily basis with the manufacturer's phantom according to manufacturer guidelines. Short-term root mean square coefficient of variation at our center is 1.1% at the lumbar spine and 1.5% at the total hip.

E2b.4. Laboratory Assays: Bone formation markers (osteocalcin, procollagen type-I N-terminal propeptide [P1NP]) and bone resorption markers (β C-terminal telopeptide of type 1 collagen [β-CTX]) correlate strongly with rates of bone formation and resorption respectively and provide powerful data as they reflect the average bone turnover globally across all bone surfaces in the body. The disadvantage of these markers is that they reflect the final state at the time of sampling and not conditions at any other time point in the experiment.

After an overnight fast, serum will be assayed from subjects between 8 and 9 am to control for diurnal variation. Blood samples will be collected and processed by nurses at the Grady GCRC core laboratory. Serum will be sent to the lab of Dr. George Beck and stored at -80◦C. The following analyses will be done at the end of the study in a single batch for each marker. Please see table 2 for details of each assay.

ELIGIBILITY:
Inclusion Criteria:Subjects with T2DM who are:

* naïve to insulin and TZD therapy
* On diet and lifestyle therapy along with submaximal metformin therapy
* with HbA1c between 7% and 8.0%
* between the ages of 18 and 80 years
* both genders

Exclusion Criteria:

* Contraindications to TZD therapy including congestive heart failure class III or IV, and/or macular edema
* history of osteoporosis (T score < -2.5 on DXA scanning) or osteoporotic fragility fracture
* treatment with glucocorticoids within 1 year of study enrollment
* treatment with bisphosphonates,calcitriol, raloxifene, Calcitonin, estrogen
* vitamin D insufficiency, defined as 25(OH)D levels <30 ng/mL or
* hyperparathyroidism
* liver disease (LFTS > 3x upper limits of normal)
* Kidney disease Cr>1.4 in females and Cr>1.5 in males
* smokers (active or within a month from stopping)
* alcohol or drug abuse/dependence
* hypogonadism in males
* mental conditions rendering the subject unable to understand the scope of the study
* female subjects who are pregnant or breast feeding
* chronic obstructive pulmonary disease
* obstructive sleep apnea.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2009-04; Primary Completion 2010-10 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Natasha B Khazai, M.D., Principal Investigator — Emory University
Locations (1):
- Grady Diabetes Clinic, Atlanta, Georgia, United States

REFERENCES:
- [Result] Beck GR Jr, Khazai NB, Bouloux GF, Camalier CE, Lin Y, Garneys LM, Siqueira J, Peng L, Pasquel F, Umpierrez D, Smiley D, Umpierrez GE. The effects of thiazolidinediones on human bone marrow stromal cell differentiation in vitro and in thiazolidinedione-treated patients with type 2 diabetes. Transl Res. 2013 Mar;161(3):145-55. doi: 10.1016/j.trsl.2012.08.006. Epub 2012 Sep 27. PMID 23022285

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 3/09 to 4/11, diabetes clinic and grady hospital
Pre-assignment Details: one participant failed to disclose that she was already on pioglitazone and was excluded
Groups:
- Pioglitazone: half of the diabetic patients will be randomized to pioglitazone treatment for 6 months starting out with 15mg qday for 4 weeks and if no adverse effects noted increased to 30mg qday for 5 more months.
- Placebo: The other half will be randomized to placebo, starting out with 15mg qday for 4 weeks and if no adverse effects noted increased to 30mg qday for 5 more months.
Period: Overall Study
Arm/Group | Pioglitazone | Placebo
Started | 5 | 5
Completed | 4 | 4
Not Completed | 1 | 1
Not completed — Adverse Event | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Pioglitazone: half of the diabetic patients will be randomized to pioglitazone treatment for 6 months.
- Placebo: The other half will be randomized to placebo.
- Total: Total of all reporting groups
Arm/Group | Pioglitazone | Placebo | Total
Number analyzed (Participants) | 5 | 5 | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 3 | 8
  >=65 years | 0 | 2 | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 52 (10) | 60 (6) | 55 (5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 7
  Male | 1 | 2 | 3
Region of Enrollment [Number; unit: participants]
  United States | 5 | 5 | 10

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Number of Osteoblast and Adipocyte Colony Forming Units Cultured From Bone Marrow Stem Cells Harvested 6 Months After Treatment With Study Drug Compared to Baseline
Description: To determine the effect of PIO (pioglitazone) on BMSC (bone marrow stem cell) lineage choice in vivo, a bone marrow aspiration was obtained from patients at baseline and after 6 months of treatment with PIO or placebo. The bone marrow was used for ex vivo CFU-OB (Colony forming units-Osteoblast) and CFU-AD assays using the same protocol described for the in vitro studies previously. We also analyzed the number of total colonies per patient at both baseline and final visit.
Time Frame: 6 months
Measure: Mean (Standard Error); unit: percent change from baseline to 6months
Groups:
- Pioglitazone-Osteoblast CFU (Colony Forming Units): Percent change in Osteoblast CFU numbers as stained with Alizarin red S at baseline and 6 months after treatment with study drug.
- Placebo-OSteoblast CFU: Percent change in Osteoblast CFU numbers as stained with Alizarin at baseline and 6 months after treatment with study drug.
- Pioglitazone-Adipocyte CFU: Percent change in adipocyte CFU numbers as stained with Oil red O at baseline and 6 months after treatment with study drug.
- Placebo-Adipocyte CFU: Percent change in adipocyte CFU numbers as stained with Oil red O, at baseline and 6 months after treatment with study drug.
Arm/Group | Pioglitazone-Osteoblast CFU (Colony Forming Units) | Placebo-OSteoblast CFU | Pioglitazone-Adipocyte CFU | Placebo-Adipocyte CFU
Number analyzed (Participants) | 5 | 3 | 5 | 3
percent change from baseline to 6months | 0 (0) | 12 (5) | 4 (4) | -7 (3)

2. Secondary Outcome: βCTX (Carboxy Terminal Collagen Crosslinks), Osteocalcin, and Adiponectin.
Time Frame: 6 months
Measure: Mean (Standard Error); unit: percent change from baseline
Groups:
- Pioglitazone-Adiponectin: serum adiponectin percent change 6 mo after study drug Rx compared to baseline.
- Placebo-Adiponectin: serum adiponectin percent change 6 mo after placebo Rx compared to baseline.
- Pioglitazone-CTX: serum CTX percent change 6 mo after pioglitazone Rx compared to baseline.
- Placebo-CTX: serum CTX percent change 6 mo after placebo Rx compared to baseline.
- Pioglitazone-OSc: serum Osteocalcin percent change 6 mo after pioglitazone Rx compared to baseline.
- Placebo - Osc: serum Osteocalcin percent change 6 mo after placebo Rx compared to baseline.
Arm/Group | Pioglitazone-Adiponectin | Placebo-Adiponectin | Pioglitazone-CTX | Placebo-CTX | Pioglitazone-OSc | Placebo - Osc
Number analyzed (Participants) | 5 | 3 | 5 | 3 | 5 | 3
percent change from baseline | 78.7 (100.2) | -0.6 (24.5) | -9.2 (36.4) | 0.2 (25.9) | 3.6 (22.1) | -5 (9.4)

3. Secondary Outcome: Bone Mineral Density
Time Frame: 6 months
Measure: Mean (Standard Error); unit: percent change from baseline to 6 months
Groups:
- Pioglitazone-Femoral Neck BMD; Pioglitazone -Lumbar Spine BMD: half of the diabetic patients will be randomized to pioglitazone treatment for 6 months.
- Placebo-Femoral Neck BMD; Placebo - Lumbar Spine BMD: The other half will be randomized to placebo.
Arm/Group | Pioglitazone-Femoral Neck BMD | Placebo-Femoral Neck BMD | Pioglitazone -Lumbar Spine BMD | Placebo - Lumbar Spine BMD
Number analyzed (Participants) | 4 | 3 | 5 | 3
percent change from baseline to 6 months | -4 (4.4) | -2.6 (6.3) | -1.1 (2.7) | 1.9 (4.2)

ADVERSE EVENTS:
Arm/Group | Pioglitazone | Placebo
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/5
Other Adverse Events (participants affected / at risk) | 0/5 | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No